CLINICAL TRIAL: NCT00770809
Title: Randomized Phase III Trial of Paclitaxel +Trastuzumab + Lapatinib Versus Paclitaxel + Trastuzumab as Neoadjuvant Treatment of HER2-Positive Primary Breast Cancer
Brief Title: Paclitaxel and Trastuzumab With or Without Lapatinib in Treating Patients With Stage II or Stage III Breast Cancer That Can Be Removed by Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01073; NCI-2009-01073 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000616648; CALGB 40601 (Other: Alliance for Clinical Trials in Oncology); CALGB-40601 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Male Breast Carcinoma; Stage IIA Breast Cancer AJCC v6 and v7; Stage IIB Breast Cancer AJCC v6 and v7; Stage IIIA Breast Cancer AJCC v7; Stage IIIB Breast Cancer AJCC v7; Stage IIIC Breast Cancer AJCC v7
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Lapatinib; Paclitaxel; Taxes; Trastuzumab; CT-P6; PF-05280014; trastuzumab biosimilar HLX02; Ogivri; Ontruzant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm I (THL) (Experimental): Patients receive trastuzumab 2 mg/kg IV over 30-90 minutes and paclitaxel 80 mg/m^2 IV over 1 hour once weekly and lapatinib ditosylate 750 mg PO once daily for 16 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lapatinib Ditosylate; Drug: Paclitaxel; Biological: Trastuzumab
- Arm II (TH) (Active Comparator): Patients receive trastuzumab 2 mg/kg IV over 30-90 minutes and paclitaxel 80 mg/m^2 IV over 1 hour once weekly for 16 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Biological: Trastuzumab
- Arm III (TL) (Experimental): Patients receive paclitaxel 80 mg/m^2 IV over 1 hour once weekly and lapatinib ditosylate 15000 mg PO once daily for 16 weeks in the absence of disease progression or unacceptable toxicity. (Discontinued as of 6-15-11)
  Interventions: Drug: Lapatinib Ditosylate; Drug: Paclitaxel

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Arm I (THL); Arm II (TH)
Drug: Lapatinib Ditosylate — Given PO
  Other Names: Tykerb
  Arms: Arm I (THL); Arm III (TL)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Trastuzumab — Given IV
  Other Names: ABP 980; ALT02; Biceltis; CANMab; CT-P06; CT-P6; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Hercessi; Herclon; Hertraz; Herwenda; Herzuma; HLX 02; HLX-02; HLX02; Kanjinti; Ogivri; Ontruzant; PF 05280014; PF-05280014; PF05280014; QL 1701; QL-1701; QL1701; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; Trastuzumab Biosimilar CT-P6; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar QL1701; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-herw; Trastuzumab-pkrb; Trastuzumab-qyyp; Trastuzumab-strf; Trastuzumab-zerc; Trazimera; Zercepac
  Arms: Arm I (THL); Arm II (TH)

SUMMARY:
This randomized phase III trial studies paclitaxel and trastuzumab with or without lapatinib to see how well they work in treating patients with stage II or stage III breast cancer that can be removed by surgery. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving paclitaxel with trastuzumab and/or lapatinib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. It is not yet known which regimen is more effective in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if the pathologic complete response (pCR) in the breast to neoadjuvant weekly paclitaxel with trastuzumab plus lapatinib (THL) is 20% greater than the pCR to weekly paclitaxel with trastuzumab alone (TH).

SECONDARY OBJECTIVES:

I. To determine the pathologic complete response in the breast and axilla, using American Joint Committee on Cancer (AJCC) Tumor, Lymph Nodes and Metastasis (TMN) criteria (version 6), to neoadjuvant weekly paclitaxel plus human epidermal growth factor 2 (HER2)- targeted therapy in patients with HER2-positive operable breast cancer.

II. To evaluate residual cancer burden (RCB) as a predictor of long term relapse free survival (RFS) and overall survival (OS).

III. To document the toxicity of all chemotherapeutic regimens (THL, TH). IV. To determine the correlation between clinical, radiographic and pathologic response.

V. To compare overall survival (OS), relapse free survival (RFS) and time to first failure (TFF) among the treatment groups.

VI. To obtain blood, fresh frozen and fixed tumor tissue to test specific hypotheses for which biomarker data exist and to evaluate biomarkers in blood, serum and tissue that are likely to influence response to and toxicity of trastuzumab alone or trastuzumab plus lapatinib, when given with paclitaxel.

VII. To determine the surgical practice patterns for breast conservation and sentinel lymphadenectomy in patients undergoing neoadjuvant chemotherapy.

VIII. To determine the radiotherapy practice patterns for post-mastectomy and regional nodal irradiation in patients undergoing neoadjuvant chemotherapy.

IX. To evaluate pharmacogenomic determinants of toxicity.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive trastuzumab IV over 30-90 minutes and paclitaxel IV over 1 hour once weekly and lapatinib ditosylate orally (PO) once daily for 16 weeks in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive trastuzumab and paclitaxel as in arm I.

ARM III: Patients receive paclitaxel and lapatinib ditosylate as in arm I. (Discontinued as of 6-15-11) Within 42 days after completion of neoadjuvant therapy, patients in both arms undergo definitive surgery (breast conservation or total mastectomy).

After completion of study treatment, patients are followed every 6 months for 2 years and then annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic confirmation of invasive breast cancer; patients with inflammatory breast cancer are not eligible
* Clinical stage II-III operable invasive breast cancer with intent to perform surgical resection after neoadjuvant therapy

  * Patients with multicentric or bilateral disease are eligible as long as the target lesion meets the eligibility criteria for this study
  * Staging to rule out metastatic disease is recommended for clinical stage III patients
* Tumors must be HER2 positive defined as HER2 3+ by immunohistochemical (IHC) assays or gene amplification by fluorescence in situ hybridization (FISH) with a ratio of >= 2 on invasive tumor
* Estrogen receptor (ER) and progesterone receptor (PgR) status must be known
* The target lesion in the breast must be >= 1 cm on physical examination or by radiographic measurement; palpable axillary adenopathy will be documented but not serve as measurable disease for the primary endpoint; patients with axillary disease only are not eligible to participate
* Patient agrees to provide pretreatment biopsies
* No prior chemotherapy, hormone therapy, biologic, or radiation therapy with therapeutic intent for this cancer
* Cardiac ejection fraction must be >= 50% by echocardiogram or multiple gated acquisition (MUGA) scan
* Eastern Cooperative Oncology Group (ECOG) (Zubrod) performance status 0-1
* Patients must not be pregnant or nursing
* Absolute neutrophil count (ANC) >= 1,000/ul
* Platelet count >= 100,000/ul
* Bilirubin =< 1.5 times upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times upper limit of normal (ULN)
* Serum beta-human chorionic gonadotropin (HCG) negative (in female patients unless status-post (s/p) hysterectomy or menopausal or no menses for 24 consecutive months); assay must have a sensitivity of at least 50 mIU/mL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2009-02-24 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Carey, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (318):
- United States (317):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Sparks Regional Medical Center, Fort Smith, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Wilma Chan Highland Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Hematology and Oncology Associates-Oakland, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Saint Helena Hospital, St. Helena, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Halifax Health Medical Center-Centers for Oncology, Daytona Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists-Gainesville Cancer Center, Gainesville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Atrium Health Navicent, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Presence Resurrection Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Franciscan Saint Francis Health-Beech Grove, Beech Grove, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Reid Health, Richmond, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - HaysMed, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at Boston Medical Center - Brighton, Brighton, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional, Milford, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Comprehensive Cancer Care PC, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Foundation Medical Partners, Nashua, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Elmhurst Hospital Center, Elmhurst, New York
  - Queens Hospital Center, Jamaica, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Garnet Health Medical Center, Middletown, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Mission Hospital, Asheville, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - UNC Rex Healthcare, Raleigh, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Clinton Memorial Hospital/Foster J Boyd Regional Cancer Center, Wilmington, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Kent Hospital, Warwick, Rhode Island
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Doctor's Hospital of Laredo, Laredo, Texas
  - Texas Tech University Health Sciences Center-Lubbock, Lubbock, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Providence Holy Family Hospital, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Saint Mary's Medical Center, Huntington, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Derived] Jaehnig EJ, Fernandez-Martinez A, Vashist TD, Holt MV, Williams L, Lei JT, Moon CI, Kim BJ, Dou Y, Zhao H, Korchina V, Gibbs RA, Muzny DM, Doddapaneni H, Perou CM, Carey LA, Robles AI, Hyslop T, Wen Y, McCart L, Krek A, Petralia F, Miles G, Kavuri SM, Gillette MA, Mani DR, Carr SA, Zhang B, Ellis MJ, Satpathy S, Anurag M. Proteogenomic analysis of the CALGB 40601 (Alliance) HER2+ breast cancer neoadjuvant trial reveals resistance biomarkers. Cell Rep Med. 2025 Jun 17;6(6):102154. doi: 10.1016/j.xcrm.2025.102154. Epub 2025 Jun 5. PMID 40480221
- [Derived] Fernandez-Martinez A, Krop IE, Hillman DW, Polley MY, Parker JS, Huebner L, Hoadley KA, Shepherd J, Tolaney S, Henry NL, Dang C, Harris L, Berry D, Hahn O, Hudis C, Winer E, Partridge A, Perou CM, Carey LA. Survival, Pathologic Response, and Genomics in CALGB 40601 (Alliance), a Neoadjuvant Phase III Trial of Paclitaxel-Trastuzumab With or Without Lapatinib in HER2-Positive Breast Cancer. J Clin Oncol. 2020 Dec 10;38(35):4184-4193. doi: 10.1200/JCO.20.01276. Epub 2020 Oct 23. PMID 33095682
- [Derived] Carey LA, Berry DA, Cirrincione CT, Barry WT, Pitcher BN, Harris LN, Ollila DW, Krop IE, Henry NL, Weckstein DJ, Anders CK, Singh B, Hoadley KA, Iglesia M, Cheang MC, Perou CM, Winer EP, Hudis CA. Molecular Heterogeneity and Response to Neoadjuvant Human Epidermal Growth Factor Receptor 2 Targeting in CALGB 40601, a Randomized Phase III Trial of Paclitaxel Plus Trastuzumab With or Without Lapatinib. J Clin Oncol. 2016 Feb 20;34(6):542-9. doi: 10.1200/JCO.2015.62.1268. Epub 2015 Nov 2. PMID 26527775
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (THL) | Arm II (TH) | Arm III (TL)
Started | 118 | 120 | 67
Completed | 101 | 110 | 44
Not Completed | 17 | 10 | 23
Not completed — Adverse Event | 9 | 1 | 12
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 3 | 7
Not completed — Progression | 2 | 2 | 0
Not completed — Complicating illness | 0 | 0 | 1
Not completed — Other Medical Reasons | 2 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (THL) | Arm II (TH) | Arm III (TL) | Total
Number analyzed (Participants) | 118 | 120 | 67 | 305
Age, Continuous [Median (Full Range); unit: years] | 48.5 [24.7 to 70.8] | 50.3 [30.2 to 75.8] | 48.3 [25.8 to 74.3] | 49.4 [24.7 to 75.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 119 | 67 | 303
  Male | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 4 | 8 | 5 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 12 | 8 | 7 | 27
  White | 95 | 97 | 51 | 243
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 4 | 5 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 118 | 120 | 67 | 305
Clinical Stage [Number; unit: participants] — The American Joint Committee on Cancer (AJCC) has designated staging by tumor, node, and metastasis (TNM) classification. Stage II participants had primary tumors 0-5 cm and no regional lymph node metastases or metastases to movable ipsilateral level I, II axillary lymph node or primary tumors > 5.1 cm and no regional lymph node metastases. Stage III participants had primary tumors of any size but not any metastases in ipsilateral infraclavicular (level III axillary) lymph node(s) with or without level I, II axillary lymph node involvement
  participants
    Stage II | 81 | 80 | 48 | 209
    Stage III | 37 | 40 | 19 | 96
Hormone Receptor Status [Number; unit: participants]
  ER/PgR Positive | 70 | 70 | 39 | 179
  ER/PgR or Negative | 48 | 50 | 28 | 126

OUTCOME MEASURES:

1. Primary Outcome: pCR Rate
Description: Complete pathological response is defined as the absence of residual invasive carcinoma in the breast at the time of definitive surgical removal. Pathologic complete response in the lymph nodes is defined as no detectable invasive tumor by H&E. Analysis will use a chi-square test for the difference in proportions of patients on the THL arm versus the TH arm who achieve a pCR. Exact binomial methods will be used to construct 95% confidence intervals around the pCR incidence for each arm.
Time Frame: At time of surgery
Population: Participants who did not start protocol therapy or withdrew prior to surgery are excluded. Participants who did not undergo surgery are considered no having a pCR.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (THL) | Arm II (TH) | Arm III (TL)
Number analyzed (Participants) | 116 | 117 | 63
percentage of participants | 56 [47 to 65] | 46 [35 to 55] | 32 [22 to 45]
Statistical Analysis 1: Comparison: Arm I (THL) vs Arm II (TH); Test type: Superiority or Other; p = 0.13, Log Rank — Participants were stratified by clinical stage (II vs III) and hormone receptor status (positive/negative)
Statistical Analysis 2: Comparison: Arm II (TH) vs Arm III (TL); Test type: Superiority or Other; p = 0.072, Log Rank — Participants were stratified by clinical stage (II vs III) and hormone receptor status (positive/negative)

2. Secondary Outcome: Pathologic Stage in the Breast and Axilla
Description: Stage will be determined by the American Joint Committee on Cancer (AJCC) TNM (tumor, lymph nodes, metastasis) staging system.
Time Frame: At time of surgery
Reporting Status: Not Posted

3. Secondary Outcome: Radiographic Response Rate (at Completion of Neoadjuvant Therapy)
Description: Response was defined by the Response Evaluation Criteria in Solid Tumors (RECIST). A responding participant had either a complete response (disappearance of all target lesions) or partial response (30% decrease in sum of longest diameter of target lesions).
Time Frame: Week 16
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival
Description: Overall survival was measured as the interval from study entry until death, from any cause, or last contact. Distribution was estimated using the Kaplan Meier product-limit method
Time Frame: Time from randomization to death or last follow-up (up to 10 years)
Reporting Status: Not Posted

5. Secondary Outcome: Relapse-free Survival (RFS)
Description: Relapse free survival is defined as the interval from definitive surgery to ipsilateral invasive breast tumor recurrence, regional invasive breast cancer recurrence, distant recurrence, or death from any cause, whichever occurs first. Patients who have not experienced any of these events will be censored at the date of last clinical assessment. Patients who do not undergo definitive surgery will not be assessable for RFS. Distribution was estimated using the Kaplan Meier product-limit method.
Time Frame: Time from surgery to any recurrence (up to 10 years)
Reporting Status: Not Posted

6. Secondary Outcome: Time to First Failure
Description: Time to first failure is defined as the interval from study entry to ipsilateral invasive breast tumor recurrence, regional invasive breast cancer recurrence, distant recurrence or death from any cause. Patients who have not experienced any of these events will be censored at the date of last clinical assessment. Distribution was estimated using the Kaplan Meier product-limit method.
Time Frame: Time from study entry to any recurrence ( up to 10 years)
Reporting Status: Not Posted

7. Secondary Outcome: Incidence of Adverse Events as Graded by the National Cancer Institute Common Terminology Criteria for Adverse Events Version 3
Description: The type and grade of treatment-related toxicity will be tabulated by treatment arm.
Time Frame: Up to 30 days post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Adverse Event data is available on 295 participants (Arm I: 115. Arm II: 115, Arm III: 65)
Arm/Group | Arm I (THL) | Arm II (TH) | Arm III (TL)
Serious Adverse Events (participants affected / at risk) | 15/115 | 12/115 | 6/65
Other Adverse Events (participants affected / at risk) | 114/115 | 114/115 | 64/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (THL) (N=115) | Arm II (TH) (N=115) | Arm III (TL) (N=65)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 9 (11) | 7 (8) | 4 (5)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 12 (16) | 5 (5) | 5 (6)
Nausea (Gastrointestinal disorders) | 7 (9) | 2 (3) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 11 (15) | 8 (9) | 4 (4)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Gallbladder infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (4) | 0 (0) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 2 (2) | 3 (3)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (3) | 1 (1) | 2 (2)
Leukocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (6) | 3 (4) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (7) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 5 (7) | 2 (3) | 4 (4)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (THL) (N=115) | Arm II (TH) (N=115) | Arm III (TL) (N=65)
Blood disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 74 (232) | 72 (218) | 40 (114)
Hemolysis (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 4 (5) | 4 (5) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Watering eyes (Eye disorders) | 0 (0) | 1 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (3) | 2 (2) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 6 (10) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 100 (307) | 55 (110) | 56 (148)
Dyspepsia (Gastrointestinal disorders) | 3 (5) | 4 (9) | 2 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 3 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 61 (136) | 45 (94) | 32 (66)
Oral hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 18 (28) | 13 (14) | 16 (23)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (3)
Edema limbs (General disorders) | 4 (5) | 6 (7) | 1 (2)
Fatigue (General disorders) | 101 (313) | 97 (319) | 47 (140)
Fever (General disorders) | 2 (2) | 1 (1) | 0 (0)
General symptom (General disorders) | 0 (0) | 1 (1) | 1 (1)
Localized edema (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 3 (6)
Hepatobiliary disease (Hepatobiliary disorders) | 0 (0) | 1 (3) | 0 (0)
Hypersensitivity (Immune system disorders) | 11 (16) | 14 (18) | 8 (9)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 2 (3) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intraoperative hepatobiliary injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 15 (26) | 9 (19) | 6 (6)
Alkaline phosphatase increased (Investigations) | 2 (4) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 12 (20) | 8 (14) | 4 (4)
Blood bilirubin increased (Investigations) | 2 (3) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 7 (11) | 6 (10) | 4 (7)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 41 (60) | 29 (51) | 19 (40)
Platelet count decreased (Investigations) | 2 (4) | 2 (4) | 3 (3)
Weight gain (Investigations) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 3 (6) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (5) | 4 (11) | 2 (6)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 8 (11) | 0 (0) | 4 (5)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 28 (49) | 34 (75) | 22 (38)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 4 (8) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 92 (229) | 84 (198) | 44 (125)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (4) | 1 (3)
Depression (Psychiatric disorders) | 1 (2) | 1 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 6 (8) | 4 (7) | 3 (3)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (6)
Irregular menstruation (Reproductive system and breast disorders) | 2 (4) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (8) | 4 (7)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (9) | 10 (23) | 1 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 5 (5) | 10 (10) | 4 (7)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (2) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 1 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 83 (243) | 49 (92) | 48 (137)
Skin disorder (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (5) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Hot flashes (Vascular disorders) | 1 (1) | 8 (12) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 4 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less